CLINICAL TRIAL: NCT02844387
Title: Oral L-arginine Supplementation in Patients With Non-resectable Brain Metastases Treated With Radiation Therapy With Palliative Intent
Brief Title: Supplementation of L-arginine in Patients With Non-resectable Brain Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Oncología Ángel H. Roffo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LABM-1
Record Dates: First submitted 2016-06-21; First posted 2016-07-26 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Unresectable Multiple Brain Metastases
Keywords: cancer; brain; arginine; radiation
MeSH Terms: conditions — Neoplasms | interventions — Arginine; N(alpha)-lauroylarginine ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arginine (Experimental): In the Arginine arm patients will receive 10 mg of L-arginine hydrochloride solution oral supplementation (in 200 ml of flavoured drinking water solution) administered twice a day prior to the radiation therapy fraction
  Interventions: Dietary Supplement: L-arginine hydrochloride solution
- Placebo (Placebo Comparator): In the Placebo arm patients will receive 200 ml of flavoured drinking water oral solution administered twice a day prior to the radiation therapy fraction
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine hydrochloride solution — Patients with unresectable brain metastases from solid tumors that are candidates from twice-daily fractionated radiation therapy will be randomized to receive either oral arginine supplementation one-hour prior to each fraction of radiation. Radiation therapy consist in whole-brain treated by two lateral fields to a total dose of 32 Gy in 20 fractions of 1.6 Gy each two times a day with a 6 hours interval between treatments (10 days), followed by a 22.4 Gy boost over the evident lesions with the same fractionation schedule (7 days). The spinal cord dose will be limited to 40 Gy
  Other Names: L-arginine; Arginine; L-arginine monohydrochloride
  Arms: Arginine
Other: Placebo — Patients with unresectable brain metastases from solid tumors that are candidates from twice-daily fractionated radiation therapy will be randomized to receive oral placebo one-hour prior to each fraction of radiation. Radiation therapy consist in whole-brain treated by two lateral fields to a total dose of 32 Gy in 20 fractions of 1.6 Gy each two times a day with a 6 hours interval between treatments (10 days), followed by a 22.4 Gy boost over the evident lesions with the same fractionation schedule (7 days). The spinal cord dose will be limited to 40 Gy
  Other Names: flavoured drinking water solution
  Arms: Placebo

SUMMARY:
This study evaluates the nutritional supplement arginine as supportive measure for patients with unresectable metastatic brain tumors that receive radiation therapy with palliative intent

DETAILED DESCRIPTION:
Brain metastasis, the most common intracranial tumor, is associated with neurological disability and short survival time. For selected patients this outcome can be improved by achieving greater local control. Virtually all cancer patients with brain metastases receive radiotherapy; a majority as part of their primary treatment while others in connection with surgery or palliation. Agents that increase the sensitivity of cancer cells to radiation may improve the control of the disease. Previous data indicates that arginine supplementation can modify the metabolism of cancer and immune cells making tumors more susceptible to standard treatments liked radiation. In this phase 1/2 comparative study the investigators will investigate whether 10 mg of arginine oral supplementation (compared to placebo administration) administered twice a day prior to the radiation therapy can modify tumor metabolism, immune response and effect of radiation. The primary end-points are safety and toxicity of arginine, quality-of-life and clinical response. The secondary end-points are imaging response and neurological progression-free survival. Additional exploratory end-points include intensity of radiation administered, effects on tumor metabolism by magnetic resonance spectroscopy, immune response by cytokine pattern in serum, body composition and nutritional parameters , overall survival and progression free survival

ELIGIBILITY:
Patients with pathology-confirmed diagnostic of solid cancer and measurable brain metastases by CT scan and/or MRI

Inclusion Criteria:

* Unresectable criteria by neurosurgeon
* Recursive partitioning analysis (RPA) -Radiation Therapy Oncology Group (RTOG) class II (Karnofsky's performance score ≥ 70 and extracranial metastases and/or non-controlled primary tumor)
* Measurable brain lesion/s by contrast-enhanced CT or MRI
* Absolute granulocyte count more or equal than 2000/mm3
* Hemoglobin more or equal than 9 g/L (patients with lower levels were transfused before the randomization)
* Normal renal laboratory (serum creatinine <1.5 mg/dL and 24-h creatinine clearance >60 mL/min)
* Normal hepatic function (aspartate aminotransferase and alanine aminotransferase <2.5 times the upper limit of normal)
* Stable body weight and composition for at least one month prior enrollment

Exclusion Criteria:

* Prior treatment for brain metastases and/or brain tumor.
* Primary brain tumor
* Hematologic malignancies
* Solid tumors of germinal origin
* Contraindication for external radiation therapy.
* Allergy to L-arginine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the scoring form NCI CTCAE v3 for detecting and quantifying potential adverse events | Baseline and thereafter every 7 days starting from day 1 of L-arginine or placebo administration and through study completion, an average of 1 year
  NCI CTCAE v3 form will be completed baseline and every 7 days starting from day 1 of L-arginine or placebo administration thereafter. This form will detect adverse events including clinical laboratory alterations associated with the administration of of L-arginine or placebo including those that may exacerbate the adverse events expected from the radiation therapy
Change from baseline of quality of life questionnaire | Baseline and thereafter every 7 days starting from day 1 of L-arginine or placebo administration and through study completion, an average of 1 year
  Quality of life questionnaire with assessment of the Karnofsky's index will be completed baseline and every 7 days starting from day 1 of L-arginine or placebo administration thereafter
Change from baseline in signs and symptoms of neurological disease | Baseline and at 4 weeks counted from the last day of treatment
  Signs and symptoms of neurological disease will be evaluated by caregiver and investigator according to response criteria evaluation guidelines. Clinical response will be considered as the changes in signs and symptoms that occur between baseline state and 30 days counted from the last day of treatment

SECONDARY OUTCOMES:
Imaging response | One month after the last day of radiation and one month after the first response assessment
  The investigators will follow the R.E.C.I.S.T. criteria for imaging and overall response evaluation
Neurological progression-free survival | Time with no radiological or symptomatic progression counted from the first of radiation therapy until the day of first documented neurological progression or date of death from any cause, whichever came first, assessed up to 50 months
  The investigators will follow the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines for imaging (CT and MRI) response evaluation based on measurable disease, assessed up to 50 months

OTHER OUTCOMES:
Intensity of radiation administered | From the first of radiation therapy through study completion, an average of 1 year
  Actual daily and total dose of radiation administered as fractional product of the planned (proposed) daily and total dose of radiation
effects on tumor metabolism by magnetic resonance spectroscopy | Before and one hour after the first dose of L-arginine (or placebo) administration without radiation therapy
  Before and one hour after the first dose of L-arginine (or placebo) administration without radiation therapy
Change from baseline in cytokine pattern in serum | Before treatment (baseline), at 4 weeks after the last of treatment and at 8 weeks after the last of treatment
  The investigators will determine levels of circulating (serum) cytokines in a sub-group of patients from both arms to determine immune effects of L-arginine.
  Comments [5] :
Change from baseline in body weight | Baseline and thereafter every 7 days starting from day 1 of L-arginine or placebo administration and through study completion, an average of 1 year
  Body weight (kg) will be determined baseline and every 7 days starting from day 1 of L-arginine or placebo administration thereafter. The reported value will be number of patients with change of 10% or higher in any value at any time point from baseline
Progression free survival | Time with no radiological or symptomatic progression in any site of disease counted from the first of radiation therapy until the day of first documented disease progression or date of death from any cause, whichever came first, assessed up to 50 months
  The investigators will follow the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines for imaging (CT and MRI) response evaluation based on measurable disease assessed up to 50 months
Overall survival | Survival time counted from the first of radiation therapy until the date of death from any cause or lost of follow-up, assessed up to 50 months
  Survival time counted from the day 1 of radiation therapy to death or lost of follow-up, assessed up to 50 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo H Navigante, MD, Phd, Principal Investigator — Instituto de Oncología Ángel H. Roffo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Castillo L, Beaumier L, Ajami AM, Young VR. Whole body nitric oxide synthesis in healthy men determined from [15N] arginine-to-[15N]citrulline labeling. Proc Natl Acad Sci U S A. 1996 Oct 15;93(21):11460-5. doi: 10.1073/pnas.93.21.11460. PMID 8876157
- [Background] Cho-Chung YS, Clair T, Bodwin JS, Berghoffer B. Growth arrest and morphological change of human breast cancer cells by dibutyryl cyclic AMP and L-arginine. Science. 1981 Oct 2;214(4516):77-9. doi: 10.1126/science.6269181.
- [Background] Bode-Boger SM, Boger RH, Galland A, Tsikas D, Frolich JC. L-arginine-induced vasodilation in healthy humans: pharmacokinetic-pharmacodynamic relationship. Br J Clin Pharmacol. 1998 Nov;46(5):489-97. doi: 10.1046/j.1365-2125.1998.00803.x. PMID 9833603
- [Background] Kang K, Shu XL, Zhong JX, Yu TT. Effect of L-arginine on immune function: a meta-analysis. Asia Pac J Clin Nutr. 2014;23(3):351-9. doi: 10.6133/apjcn.2014.23.3.09. PMID 25164444
- [Background] Cerchietti LC, Bonomi MR, Navigante AH, Castro MA, Cabalar ME, Roth BM. Phase I/II study of selective cyclooxygenase-2 inhibitor celecoxib as a radiation sensitizer in patients with unresectable brain metastases. J Neurooncol. 2005 Jan;71(1):73-81. doi: 10.1007/s11060-004-9179-x. PMID 15719279